CLINICAL TRIAL: NCT04942288
Title: The Effect of Acupressure and Massage on the Paın, Menstrual Symptoms and Qualıty of Lıfe ın Prımary Dysmenorrhea
Brief Title: The Effect of Acupressure and Massage on Pain in Primary Dysmenorrhea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, SEDA ERYILMAZ, Principal Investigator, Inonu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020-638
Record Dates: First submitted 2021-05-19; First posted 2021-06-28 (Actual); Last update posted 2021-06-28 (Actual); Status verified 2021-06

CONDITIONS: Acupressure
Keywords: Primary Dysmenorrhea; Acupressure; Massage; Midwife
MeSH Terms: interventions — Massage

STUDY DESIGN:
Intervention Model Description: It consists of 3 Different Groups.
Masking Description: Double Blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Acupressure + Massage Group (Experimental): Acupressure + Massage Group First menstrual cycle - On the first day, Personal Information Form, VAS, GMSSS and Quality of Life Scale Short Form SF- 12 will be applied. On the first day, intervention will be made and VAS will be applied after the intervention. On the second day, VAS will be applied before and after the intervention. On the third day, VAS before and after the intervention VAS, GMSSS will be applied.
  Second menstrual cycle
  - On the first day, VAS will be applied before the intervention, and VAS will be applied after (1 hour). On the second day, VAS will be applied before and after the intervention (1st hour). On the third day, VAS before and after the intervention (1st hour) VAS, GMSSS will be applied.
  Interventions: Other: The first group is acupressure and massage, the second group is massage
- Massage Group (Experimental): Massage Group First menstrual cycle - On the first day, Personal Information Form, VAS, GMSSS and Quality of Life Scale Short Form SF- 12 will be applied. On the first day, intervention will be made and VAS will be applied after the intervention (1st hour). On the second day, VAS will be applied before and after the intervention (1st hour). On the third day, VAS before and after the intervention (1st hour) VAS, GMSSS will be applied.
  Second menstrual cycle
  - On the first day, VAS will be applied before the intervention, and VAS will be applied after (1 hour). On the second day, VAS will be applied before and after the intervention (1st hour). On the third day, VAS before and after the intervention (1st hour) VAS, GMSSS will be applied.
  Interventions: Other: The first group is acupressure and massage, the second group is massage
- Control Group (No Intervention): Control Group First menstrual cycle
  - On the first day, Personal Information Form, VAS, GMSSS and Quality of Life Scale Short Form SF-36 will be applied. On the second day, VAS will be applied. On the third day, VAS, GMSSS will be applied.
  Second menstrual cycle - On the first day, VAS, GMSSS will be applied. On the second day, VAS will be applied. On the third day, VAS, GMSSS will be applied.
  Third menstrual cycle
  - On the first day, VAS, GMSSS will be applied. On the second day, VAS will be applied. On the third day, VAS, GMSSS and Quality of Life Scale Short Form SF-12 will be applied.

INTERVENTIONS:
Other: The first group is acupressure and massage, the second group is massage — In the study, acupressure + massage will be applied to one group during 3 menstrual cycles and in the first 3 of the menstrual cycles, and only to the other group by the researcher in the experiment groups with dysmenorrhea.
  Arms: Acupressure + Massage Group; Massage Group

SUMMARY:
Painful menstrual bleeding, also known as dysmenorrhea, is one of the common gynecological ailments that have health, social, and economic implications. Dysmenorrhea has psychological effects as well as its physiological effects on women. While it negatively affects the quality of daily life and performance of women, it also causes loss in work and school life. Acupressure application has a soothing, psychological and analgesic effect. Acupressure application is also effective in reducing labor pain, low back pain, dysmenorrhea, head, neck and shoulder pain. It is thought that acupressin used in combination with pharmacological methods may be effective in relieving pain or decreasing its severity, the rate of analgesic use may be reduced, therefore analgesic side effects may be less and the patient's quality of life will increase. positively affected. It is an important part of midwifery care in terms of its application areas and benefits. As it is an effective method, it is recommended to be used in the midwifery field in the literature, it is taught and applicable, does not require medical equipment, equipment and cost. There are no studies in the literature in which non-pharmacological methods of acupressure and massage are used in primary dysmenorrhea. It is among the duties, powers and responsibilities of midwives to comfort their patients with non-invasive interventional practice. Based on these, it is thought that the use of acupressure and massage in primary dysmenorrhea is necessary to examine the level of pain, menstrual symptoms and their effects on quality of life. The type of the study was planned as a randomized controlled pre-test-post-test study. The population of the study will be students who study at Kırşehir Ahi Evran University Faculty of Education, have dysmenorrhea and meet the study criteria. In the power analysis used to determine the sample size, 5% error level and 90% power were determined as a minimum of 89 people for each group. The data of the study will be collected between December and May 2020 with the Personal Information Form in which socio-demographic characteristics are questioned, the Visual Analogue Scale for the assessment of dysmenorrhea pain, the Daily Menstrual Symptom Assessment Scale, and the Short Form of the Quality of Life Scale. (SF-12). Students who meet the inclusion criteria will be randomly selected for the experimental and control groups.

DETAILED DESCRIPTION:
Purpose of the Research:

The aim of the study is to determine the effect of acupressure and massage on pain severity, menstrual symptoms and quality of life in students with primary dysmenorrhea.

Research Hypotheses:

H1: Students who have been treated with acupressure and massage in dysmenorrhea have lower pain levels than the control group.

H2: Pain levels of students who have been treated with acupressure and massage in dysmenorrhea are lower than those who have only been massaged.

H3: The menstrual symptom intensity of students undergoing acupressure and massage in dysmenorrhea is lower than in the control group.

H4: In menstrual symptom intensity of students who have been treated with acupressure and massage in dysmenorrhea is lower than those who have been massaged only.

H5: The quality of life of students undergoing acupressure and massage in dysmenorrhea is higher than the control group.

H6: The quality of life of students who have been treated with acupressure and massage in dysmenorrhea is higher than those who have been massaged only.

Materıal Method

Type of the Study The research was planned as a randomized controlled trial.

Place and Time of the Study The research will be carried out between September 2020 and June 2021 in the Faculty of Education randomly selected among the faculties located on the campus of Kırşehir Ahi Evran University. There are 7 departments in the Faculty of Education: computer and instructional technology education, educational sciences, mathematics and science education, turkish and social sciences education, basic education, special education, foreign language education. As of 2019-2020 academic year, the total number of female students in the faculty is 1574. There is no course in the curriculum of the departments of the faculty that includes dismenor, including health information lessons.

The Universe and the Sample of the Research The universe of the research will be female students studying at the Education Faculty of Kırşehir Ahi Evran University (N = 1574). The sample of the research will be students who study at Kırşehir Ahi Evran University Faculty of Education, experience dysmenorrhea and have criteria for recruitment. For the power analysis of the study, based on the fact that Uçar et al. (2018) had a mean score of 7.44 (Standard deviation 2.0) in university students experiencing primary dysmenorrhea, assuming that the intensity of pain would be 6.6 points in 95% confidence interval, with 80% strength. the size was determined to be at least 89 for each group. (89 acupressure + massage group, 89 massage group, 89 control groups). The number of students to be taken from the departments in the faculty will be determined by proportioning the weights of the departments in the universe. For this, the number of students in each department will be requested from the faculty. Then, the Random Integer Generator method will be used to separate the experimental and control groups. For this, 267 students will be listed, and students from 3 columns in random.org will be divided into groups according to their numbers.

In the study, dysmenorrhea was defined as the pain during menstrual bleeding. The criteria included in the scope of pain in dysmenorrhea are pain in the waist, groin or abdomen that started in the first 6-12 hours and lasted for 8-72 hours in the last 12 months (Ambresin et al., 2012).

Data Collection Tools Personal Information Form (Appendix-1) in collecting data, Visual Analogue Scale (VAS) (Appendix-2), Daily Menstrual Symptom Evaluation Scale (Appendix-3), Quality of Life Scale Short Form SF-12 (Appendix-4) in the evaluation of dysmenorrhea pain It will be used.

Personal Information Form (Annex-1) The questions in the form were prepared by the researcher in line with the literature information. In this form, students; The questions questioning the characteristics (age, department, number of class), and the features associated with the menstrual cycle (age of menarche, bleeding time, pain duration, etc.) were included.

Visual Analog Scale (VAS) (Annex-2) VAS is used to measure perceived pain. Painlessness on one end and 10 cm on the other for the most severe pain. On a (100 mm.) Ruler, the patient expresses his pain by drawing a line, marking or pointing. The length of the distance from where there is no pain to the point marked by the patient is measured in centimeters, and the numerical value found indicates the pain intensity of the patient.

Daily Menstrual Symptom Evaluation Scale (GMSSS) (Annex-3) GMSSS was developed by Jenni W. Taylor (1979) to evaluate the symptoms and intensity of symptoms that occurred during menstruation. The Turkish validity and reliability of the scale was performed by Oskay et al. The intensity of each symptom is scored between 0 and 5 on a scale of 17 symptoms. Increased score indicates that the intensity of symptoms increases. In the study of Oskay et al. (2008), Cronbach's alpha value of the scale was found to be 0.88.

Quality of Life Scale Short Form SF-12 (Annex-4) A shorter form SF-12 Short Health Scale was created by taking 12 different items from 8 different subtitles of SF-36.

SF-12 has a physical (SF12-PCS) and mental (SF12-MCS) status assessment scale with regression analysis applied in the general population. SF-12 was developed and version 2.0 (SF-12v2) was created. Words are shortened and simplified, questions and answers are made easier to read to prevent missing answers, 6-step answer categories are reduced to 5 by reducing complexity, and answers are simplified by printing in a horizontal (left to right) form.

SF-12 is an easy-to-apply survey, obtained by shortening and simplifying SF-36, with proven reliability and validity. It is used in the evaluation of physical and mental health, which are two main components of general health status.

The T-score used when calculating scoring in SF-36 is not used in SF-12. Instead, it is not possible to calculate if there is missing data in SF-12, which has a different scoring rule.

Research Variables Independent Variables: Acupressure and massage treatments applied to students experiencing dysmenorrhoea Dependent Variables: Pain severity, menstrual symptoms, quality of life levels of students experiencing dysmenorrhea

ELIGIBILITY:
Inclusion Criteria:

* Having a regular messtruation period (lasting 3-8 days, 21-35 days in the menstrual cycle),
* Dismenorrhea pain intensity is 4 and over according to VAS,
* Do not use any medication at least 8 hours before the intervention.

Exclusion Criteria:

* Diagnosed with secondary dysmenorrhea (endometriosis, ovarian cyst / tumor, pelvic infection disease, myoma, uterus polyp, uterus adhesions, infection)
* Using oral contraceptives,
* Disruption of tissue integrity in the abdominal region,
* Any chronic or mental illness.

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — A study we will do during the menstruation period of female students
Enrollment: 267 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2020-12-12 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Pain in Primary Dysmenorrhea | Change in pain after three months
  The VAS scale was used to measure pain. The VAS scale is 10 cm, with painlessness at one end and the most severe pain at the other. On a (100 mm.) ruler, the patient describes his or her pain by drawing a line, pointing, or pointing. The distance from the point where there is no pain to the point marked by the patient is measured in centimeters and the numerical value found indicates the severity of the patient's pain.

SECONDARY OUTCOMES:
Quality of Life Scale | Change in quality of life after three months
  SF-12 was used to assess quality of life. In the calculation, physical standardization values and mental standardization values are collected separately. The summary of the physical components is calculated by adding 56.57706 to the total of physical standardization for 12 questions, and the summary of mental components is calculated by adding 60,75781 to the total of mental standardization for 12 questions. High scores indicate good health.
Daily Menstrual Symptom Rating Scale | Change in menstrual symptom intensity after three months
  Daily Menstrual Symptom Rating Scale (GMSS) was used. The intensity of each symptom is scored between 0 and 5 on a 17-symptom scale. An increase in score indicates an increased intensity of symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Seda ERYILMAZ, Msc, Principal Investigator — Kirsehir Ahi Evran Universitesi
Locations (1):
- Faculty of Health Science, Kırşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
İndividual participant data were not shared

REFERENCES:
- [Background] Chen HM, Chen CH. Effects of acupressure on menstrual distress in adolescent girls: a comparison between Hegu-Sanyinjiao matched points and Hegu, Zusanli single point. J Clin Nurs. 2010 Apr;19(7-8):998-1007. doi: 10.1111/j.1365-2702.2009.02872.x. PMID 20492044
- [Result] Wong CL, Lai KY, Tse HM. Effects of SP6 acupressure on pain and menstrual distress in young women with dysmenorrhea. Complement Ther Clin Pract. 2010 May;16(2):64-9. doi: 10.1016/j.ctcp.2009.10.002. Epub 2009 Nov 14. PMID 20347835
- [Derived] Eryilmaz S, Ucar T. The Effects of Acupressure and Massage on Pain, Menstrual Symptoms, and Quality of Life in Primary Dysmenorrhea: A Randomized Controlled Trial. J Integr Complement Med. 2025 Apr;31(4):378-387. doi: 10.1089/jicm.2023.0721. Epub 2024 Dec 20. PMID 39705091